CLINICAL TRIAL: NCT01345799
Title: A Two Part, Multi-Centre, Randomized, Placebo-Controlled, Double-Blind Study of TRK-170 for the Treatment of Crohn's Disease
Brief Title: A Study of TRK-170 for the Treatment of Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 170CDT01
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease Activity Index; Crohn's Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- TRK-170 Low Dose (Experimental)
  Interventions: Drug: TRK-170
- TRK-170 Middle Dose (Experimental)
  Interventions: Drug: TRK-170
- TRK-170 High Dose (Experimental)
  Interventions: Drug: TRK-170
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRK-170
  Arms: TRK-170 High Dose; TRK-170 Low Dose; TRK-170 Middle Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
In Crohn's Disease Patients

* To evaluate the efficacy of TRK-170
* To evaluate the PK characteristics of TRK-170
* To assess the safety of TRK-170

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of Crohn's Disease before screening
* Patient has stable disease activity

Exclusion Criteria:

* Patient has had a clinically significant illness prior to screening
* Patient with clinically significant deviations in laboratory values

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2011-04; Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index | 12 weeks
  8 weeks (treatment), 4 weeks (follow-up)

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium, Belgium, Belgium
- Bulgaria, Bulgaria, Bulgaria
- Czech Republic, Czech Republic, Czechia
- France, France, France
- Hungary, Hungary, Hungary
- Latvia, Latvia, Latvia
- The Netherlands, The Netherlands, Netherlands
- Norway, Norway, Norway
- Poland, Poland, Poland
- Romania, Romania, Romania
- Serbia, Serbica, Serbia
- Sweden, Sweden, Sweden
- Ukraine, Ukraine, Ukraine